CLINICAL TRIAL: NCT01972958
Title: Effects of Community Health Programs by Nurses for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200908042R
Record Dates: First submitted 2013-10-18; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Older Adults
MeSH Terms: interventions — Comprehensive Health Care; Community Health Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- comprehensive care (Experimental): comprehensive assessment, physical activity training, community resources referral, health education, health promotion activity.
  Interventions: Other: comprehensive care
- usual care (No Intervention): control group with usual care

INTERVENTIONS:
Other: comprehensive care — comprehensice assessment,physical activity training, community resources referral, health education.
  Other Names: community health care
  Arms: comprehensive care

SUMMARY:
As the aging population increases, preventing and decreasing disabilities become a critical issue for the health care system. Previous researches have shown that preventive community-based nursing services for older adults could achieve important health benefits at a relatively low cost. However, many frail and pre-frail older adults living in communities cannot get enough attention from current health care system. The role and function of nurses should be expanded to provide more comprehensive family-oriented care to improve health outcomes of older adults in Taiwan. The objectives of this study are:

1. Understand the difficulties and solutions for nurses providing community-based services in order to expand their better role and function.
2. Develop a cultural sensitive community advanced nurse service model for Taiwan in health care system.
3. Explore the effectiveness of community health programs by nurses for frail or pre-frail older adults in community.

Focus groups and literature review will be used to achieve the first and second study objectives. A single centre randomized controlled trial will be used in this study to achieve the third study objective. Two hundred and twenty people aged 65 and over who meet the Fried definition of frailty and pre-frailty will be recruited from the clinic of a hospital. Participants will be followed for a 6-month period. Frailty, quality of life, satisfaction to the services, hospitalizations and admissions to nursing care facilities will be measured and compared between experimental group and control group. This research is an important step in the examination of a new approach to the community older people by nurses. The study results will provide the evidence data to recommendation for related policy making in the future.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and above, frail and pre-frail older adults, living in communities

Exclusion Criteria:

* Cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lian-Hua Huang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School of Nursing, National Taiwan University, Taipei, Taiwan, Taiwan